CLINICAL TRIAL: NCT06297772
Title: Comparing the Efficacy and Safety of Decitabine-Fludarabine-busulfan (Dec-FB4) and Fludarabine-busulfan (FB4) as Conditioning Regimens for AML-MR
Brief Title: Compare the Efficacy and Safety of Dec-FB4 and FB4 as Conditioning Regimen for AML-MR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Xiaoxia, Principal Investigator, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJBMT-003
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: AML, Adult
Keywords: AML-MR; adults; conditioning regimen
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; fludarabine; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flu-Bu4 (Active Comparator): Preconditioning with Flu-Bu4 without decitabine for patients with AML-MR
  Interventions: Drug: Fludarabine Injection; Drug: Busulfan Injection
- Dec-Flu-Bu4 (Experimental): Preconditioning with Flu-Bu4 and decitabine for patients with AML-MR
  Interventions: Drug: Decitabine; Drug: Fludarabine Injection; Drug: Busulfan Injection

INTERVENTIONS:
Drug: Decitabine — decitabine 20mg/m2 per day for consecutive 5 days
  Arms: Dec-Flu-Bu4
Drug: Fludarabine Injection — fludarabine 30mg/m2 per day for consecutive 5 days
Drug: Busulfan Injection — Busulfan 3.2mg/kg per day for consecutive 4 days

SUMMARY:
A multicenter, randomized, controlled clinical study comparing the efficacy and safety of allogeneic hematopoietic stem cell transplantation with decitabine-Fludarabine- busulfan (Dec-FB4) and Fludarabine-busulfan (FB4) as pretreatment regimens for the treatment of acute myeloid leukemia in adults with MR gene abnormalities

DETAILED DESCRIPTION:
AML-MR is one of high-risk AML with aggressive disease progression and poor prognosis. The median survival of AML-MR is only 10.5 months. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective post-remission therapy for high-risk acute myeloid leukemia (AML)/myelodysplastic syndrome (MDS). Selection of an appropriate pretreatment regimen that balances the risk of relapse and reduces the risk of non-relapse mortality is a key component of successful HSCT. FB4 regimen consisting of Fludarabine (FLU) combined with busulfan (BU) has become the most commonly used myeloablative preconditioning regimen for allo-HSCT in patients with AML/MDS, and prospective studies have demonstrated a similar relapse rate and lower treatment-related mortality than the Bu/cy regimen.

Decitabine is also approved for the treatment of AML and MDS as an inhibitor of DNA methyltransferase I, which allows for the expression of silenced oncogenes and terminal differentiation of leukemia cells, and as a single agent is superior to supportive therapy for patients with MDS. In addition, decitabine has been shown to attenuate GVHD by enhancing the function of regulatory T cells, and in myeloid tumors, several prospective single-arm and retrospective clinical studies have demonstrated that modified pretreatment regimens containing decitabine have a lower relapse rate, as well as a reduction in the incidence and severity of GVHD, with satisfactory survival data in allogeneic hematopoietic stem cell transplantation. The investigators have not yet obtained direct evidence in high-risk patients to confirm the superiority of decitabine-containing pretreatment regimens over standard pretreatment regimens (FB4). There is a lack of prospective, controlled studies to clarify the efficacy and safety of decitabine-containing transplantation preconditioning in high-risk patients, especially those with specific AML-MR.Therefore, this multicenter, randomized controlled study was designed to compare the efficacy and safety of Dec-FB4 and FB4 regimens as pretreatment regimens for allogeneic HSCT in adults with AML-MR and to assess whether Dec-FB4 is superior or noninferior to FB4, in order to provide a reliable evidence-based medical basis for guiding the therapeutic choices for AML-MR/MDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-65 years and with an ECOG physical fitness score of 0-2 and an HCT-CI of less than 3;
* Diagnosis: All enrolled cases were diagnosed with acute myeloid leukemia (AML-MR) after bone marrow cytomorphology, cytochemistry, immunophenotyping, chromosomal examination, and gene mutation, and achieved hematological remission (bone marrow smear primitive cells <5%) and negative MRD before transplantation.
* Have a medically qualified and suitable hematopoietic stem cell donor, including HLA-allogamous sibling donors, unrelated donors (HLA high-resolution 9-10/10 compatible) or related haploidentical donors;
* No dysfunction of the heart, liver, lungs, kidneys, or other important organs, as defined as follows: ALT and AST ≤3 times the upper limit of normal; total bilirubin ≤2 times the upper limit of normal); BUN and Cr ≤1.25 times the upper limit of normal; electrocardiograms not suggestive of acute myocardial infarction or serious arrhythmias; cardiac echocardiography left ventricular ejection fraction ≥50%, no significant cardiac enlargement, valvular disease, or congenital heart disease; pulmonary function examination FEV1, FVC, DLCO ≥ 60% of the predicted value.
* The patient and his/her legal representative have the desire and requirement to undergo hematopoietic stem cell transplantation and sign an informed consent, willingness and compliance with the treatment plan, follow-up schedule, laboratory tests, etc.

Exclusion Criteria:

* AML in unremitting stage; or BM in remission but with concurrent CNS leukemia or presence of extramedullary lesions;
* Active hepatitis B (HBV-DNA ≥1×10^3 copies/ml);
* HIV-infected patients;
* Active infections requiring intravenous antibiotic therapy;
* There is severe impairment of vital organ function: respiratory failure, heart failure, decompensated hepatic insufficiency, renal insufficiency, etc;
* Patients who use drugs or chronic alcohol abuse to the extent that it interferes with the evaluation of test results;
* Mentally challenged/unable to obtain informed consent;
* Those judged by the investigator to be unsuitable for participation in this trial.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | through study completion, an average of 2 year
  disease progression or death as a result of any causes

SECONDARY OUTCOMES:
incidence of relapse rate | through study completion, an average of 2 year
  disease relapse
Non-recurrent mortality | through study completion, an average of 2 year
  death without disease progression or relapse

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxia Hu, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, China